CLINICAL TRIAL: NCT04791956
Title: Double-blind, Randomized Placebo-controlled Trial Investigating the Effect of Prebiotic Inulin-type Fructans on Bowel Habits of Infants
Brief Title: Prebiotic EffecT InfanTs
Acronym: PETIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beneo-Institute (Industry)
Collaborators: Hospital Universitari Sant Joan de Reus (Other); Hospital de Tarragona Joan XXIII (Unknown); Institut Investigacio Sanitaria Pere Virgili (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20018m-jhr
Record Dates: First submitted 2021-03-05; First posted 2021-03-10 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Infant Development; Healthy; Diet, Healthy
Keywords: Microbiota, gastrointestinal health
MeSH Terms: interventions — Prebiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prebiotic (Experimental): Inulin-type fructans
  Interventions: Dietary Supplement: Prebiotic
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Prebiotic — Daily intake of Inulin-type fructans from chicory
  Arms: Prebiotic
Dietary Supplement: Placebo — Daily intake of maltodextrin
  Arms: Placebo

SUMMARY:
The study aims to confirm the effectiveness of chicory-derived prebiotic inulin-type fructans on stool consistency in infants.

DETAILED DESCRIPTION:
The fermentation of prebiotic inulin-type fructans leads to a modulation of the gut microbiota composition, in particular to a growth stimulation of bifidobacteria, and the production of organic acids like lactate and short-chain fatty acids (SCFA). The introduction of solid foods is frequently associated with harder stools which are more difficult to pass and can cause painful defecations. Subsequently, the changes in bowel habits associated with weaning and the introduction of complementary foods could be minimized by the addition of prebiotics to complementary foods and, thus, the transition from milk-feeding to family food could be facilitated.

ELIGIBILITY:
Inclusion Criteria:

* Child is healthy at the time of pre-examination
* Child was born on term or preterm (≥ 32 weeks of gestation)
* Child is aged 6-12 months at the time of pre-examination (for preterm born children (32-37 weeks of gestation), corrected age will be applied)
* Normal growth (weight and length for age between 10th and 90th percentiles, Fenton and Kim 2013)
* Child receives at least one meal per day as complementary feeding
* Child and legal guardian are able and willing to follow the study instructions
* Child is suitable for participation in the study according to the investigator/physician/study personnel
* Written informed consent is given by parent or legal guardian

Exclusion Criteria:

* No legal guardian's command of any local language
* Organic causes of defecation disorders incl. Hirschsprung disease, Spina bifida, hypothyroidism etc.
* Other metabolic or renal abnormalities or psychomotor retardation (e.g. hypotonia)
* Child has allergy to cow's milk protein or lactose intolerance
* Child has been or is currently breast-fed more than once daily (6 weeks before intervention)
* Child has mostly loose or watery stools in ≥ 50% of defecations
* Use of drugs (e.g. antibiotics) influencing gastrointestinal function (6 weeks before intervention)
* Use of laxatives or pre- or probiotic supplements in the previous 4 weeks before intervention
* Child is currently involved or will be involved in another clinical or food study

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Stool consistency | 4 weeks
  Assessed by the parents in a continuous daily bowel diary over the study period

SECONDARY OUTCOMES:
Stool frequency | 4 weeks
  Assessed by daily parental reporting
Stool colour | 4 weeks
  Assessed by the parents in a continuous daily bowel diary over the study period
Stool amount | 4 weeks
  Assessed by the parents in a continuous daily bowel diary over the study period
Sleep | 4 weeks
  Change in sleep behavior assessed by parental questionnaire (Brief Infant Sleep Questionnaire) at the beginning and end of the trial
Stool pH | 4 weeks
  change in stool pH over a four week period
stool short-chain fatty acids | 4 weeks
  change in amount and relative distribution of short-chain fatty acids in stool over a four week period
Tolerance and acceptability | 4 weeks
  Tolerance and acceptability of the study products assessed by customized parental questionnaire at the end of the trial
Body weight | 4 weeks
  changes in body weight (kg) assessed by an investigator
Body height | 4 weeks
  changes in body height (m) assessed by an investigator
Faecal Microbiota | 4 weeks
  Stool samples will be analysed by appropriate molecular biological methods like 16S rRNA gene sequencing to gain insight into the composition of the gut microbiota.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Closa Monasterolo, Phd, MD, Principal Investigator — Paediatrics Unit, University Hospital Joan XXIII, Tarragona, Spain. Paediatrics Research Unit on Nutrition and Human Development, Universitat Rovira i Virgili, Reus, Spain; Joaquin Escribano Subias, PhD, MD, Principal Investigator — Paediatrics Unit, University Hospital Sant Joan, Reus, Spain. Paediatrics Research Unit on Nutrition and Human Development, Universitat Rovira i Virgili, Reus, Spain
Locations (2):
- Spain (2):
  - Hospital Universitari Sant Joan de Reus - Magatzem, Reus
  - Hospital Universitari Joan XXIII de Tarragona - Almacén general, Tarragona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Closa-Monasterolo R, Ferre N, Castillejo-DeVillasante G, Luque V, Gispert-Llaurado M, Zaragoza-Jordana M, Theis S, Escribano J. The use of inulin-type fructans improves stool consistency in constipated children. A randomised clinical trial: pilot study. Int J Food Sci Nutr. 2017 Aug;68(5):587-594. doi: 10.1080/09637486.2016.1263605. Epub 2016 Dec 8. PMID 27931142